CLINICAL TRIAL: NCT03567330
Title: African American Families Fighting Parental Cancer Together
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient patients meet eligibility requirements.
Sponsor: University of Delaware (Other)
Collaborators: Helen F. Graham Cancer Center & Research Institute at Christiana Care (Unknown); Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Adam Davey, Professor, Behavioral Health and Nutrition, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1165185-1
Record Dates: First submitted 2018-05-23; First posted 2018-06-25 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Depressive Symptoms; Anxiety; Parental Stress
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Group (cluster) randomized trial. Total number of participants is 200, including 100 men and 100 women.
Who Masked: Outcomes Assessor
Masking Description: Assessors and analysts will be blinded to treatment condition. Participants and providers cannot be effectively blinded to treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Family-based attachment-focused intervention for families where parent/caregiver is within 12 months of first diagnosis of a stage I-III solid tumor cancer.
  Interventions: Behavioral: Family-based attachment-focused intervention
- Psychoeducation (Active Comparator): Provides equivalent number of American Cancer Society psychoeducational sessions.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Family-based attachment-focused intervention — 5 2-hour biweekly sessions involving parent and/or adolescent(s).
  Arms: Experimental
Behavioral: Psychoeducation — Provides equivalent number of American Cancer Society psychoeducational sessions involving only parents.
  Arms: Psychoeducation

SUMMARY:
The purpose of this study is to test the usefulness of a family-based program for African American parents/primary caregivers with newly diagnosed solid tumor cancer and their adolescent children. The program is designed to promote family communication reduce and depressive symptoms for adolescence.

DETAILED DESCRIPTION:
The investigators will offer a 8-week prevention program to help African American parents and caregivers (e.g., grandparents) diagnosed for the first time with Stages 0, I, II, or III solid tumor cancer or hematologic cancer in the last 24 months who are caring for a 11-21 year old child at home who has been told about the parent's cancer diagnosis. Parents and their adolescent child(ren) will first be asked to complete a set of questionnaires that takes about 60 minutes and then will be told within 2 to 4 weeks whether they have been assigned to 1 of 2 programs that will get chosen by chance, like flipping a coin. Neither the families nor the researchers will choose what program is assigned. Both programs are designed to offer help coping with cancer. Both short- and long-term effects of the program will be evaluated.

Program A involves just parents attending five educational sessions every other week (1 hour/session) with a group of parents who are also coping with cancer with specially trained group leaders. Adolescent children will not participate in these group sessions; this is the treatment as usual comparison group as most cancer centers do not meet with adolescent children who have parents diagnosed with cancer.

Program B involves five group sessions (2 hours/session) every other week with other families like them that include adolescents in some of the sessions and parents and adolescents together in other sessions with specially trained group leaders.

The primary, secondary, and exploratory aims of this research are:

Primary Aim:

Aim 1. Compare the efficacy of Families Fighting Cancer Together (FFCT) to Treatment-as-Usual (TAU) in reducing depressive symptoms (CDI) in AA adolescents at post-treatment using an intention-to-treat (ITT) analysis.

Secondary Aim:

Aim 2. Compare the efficacy of Families Fighting Cancer Together (FFCT) to Treatment-as-Usual (TAU) in reducing parental stress (PCQ) in AA parents at post-treatment using ITT analysis.

Exploratory Aims:

Aim 3a. Determine trajectories of adolescent depressive symptoms (CDI), anxiety (RCMAS), and parental stress (PCQ) from baseline to 12-month follow-up.

Aim 3b. Determine whether perceived levels of group support (HGE), adolescent gender and age, parent's marital and socioeconomic status, and parent's cancer staging modify the effects of treatment on adolescent depression (CDI) and anxiety (RCMAS).

Aim 3c. Determine whether pre-post changes in parent-adolescent attachment and communication mediate the association between treatment and adolescent depressive symptoms (CDI) and anxiety (RCMAS) at 6- and 12-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Parents must identify as non-Hispanic Black
* Must be diagnosed for the first time with stage 0, I, II, or III solid tumor cancer (e.g., breast, prostate, colorectal, lung) or hematologic cancer in the last 24 months
* Must be parent or primary caregiver of at least 1 adolescent living (target child) at home (ages 11-21) who has been told about the diagnosis

Exclusion Criteria:

* Parents with serious mental health illness that prevents them from participating in the group sessions (e.g., clinically relevant depressive symptomatology as evidenced by the Center for Epidemiological Studies Depression Scale >27)
* Parents with psychotic features or severe cognitive impairment
* Parents not fluent in English.
* Severely depressed adolescents (CDI-2; T-scores of 70 and higher on the total 28-item CDI-2 scale
* Severely anxious adolescents (RCMAS-2; We will use a cutoff score of 71 (T-score) or higher to screen out African American adolescents with severe anxiety) at baseline
* Adolescents with psychotic features
* Adolescents with cognitive impairment (e.g., mental retardation, severe developmental disorders) as evidenced by educational records, parental report and/or clinical impression
* Adolescents currently in active outpatient mental health treatment.

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Reduce 8-week depressive symptoms among African American adolescents on the Child Depression Inventory (CDI-2) | Baseline to 8 weeks (end of treatment)
  Compare the efficacy of Families Fighting Cancer Together (FFCT) to Psychoeducation (PED) in reducing Child Depression Inventory symptoms (CDI-2) in AA adolescents at post-treatment using an intention-to-treat (ITT) analysis.

SECONDARY OUTCOMES:
Reduce 8-week parental stress among African American parents on the Parenting Concerns Questionnaire (PCQ) | Baseline to 8 weeks (end of treatment)
  Compare the efficacy of Families Fighting Cancer Together (FFCT) to Psychoeducation (PED) in reducing parenting stress on the Parenting Concerns Questionnaire (PCQ) in AA parents at post-treatment using ITT analysis.

OTHER OUTCOMES:
Reduce depressive symptoms among African American adolescents on the Child Depression Inventory (CDI-2) | Baseline to 12 months
  Compare the efficacy of Families Fighting Cancer Together (FFCT) to Psychoeducation (PED) in reducing Child Depression Inventory (CDI-2) symptoms in AA adolescents at 12 months using an intention-to-treat (ITT) analysis.
Reduce depressive symptoms among African American adolescents on the Revised Children's Manifest Anxiety Scale (RCMAS-2) | Baseline to 12 months
  Compare the efficacy of Families Fighting Cancer Together (FFCT) to Psychoeducation (PED) in reducing anxiety on the Revised Children's Manifest Anxiety Scale (RCMAS-2) in AA adolescents at 12 months using an intention-to-treat (ITT) analysis.
Reduce 8-week parental stress among African American parents on the Parenting Concerns Questionnaire (PCQ) | Baseline to 12 months
  Compare the efficacy of Families Fighting Cancer Together (FFCT) to Psychoeducation (PED) in reducing parental stress on the Parenting Concerns Questionnaire (PCQ) in AA parents at 12 months using ITT analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Davey, Ph.D., Principal Investigator — University of Delaware
Locations (2):
- United States (2):
  - Helen F Graham Cancer Center & Research Institute at Christiana Care, Newark, Delaware
  - Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- [Result] McKinney NS, Virtue S, Lewis FM, Willis AI, Pettyjohn T, Harmon LR, Davey A. Study protocol: a randomized control trial of African American families fighting parental cancer together. BMC Cancer. 2018 Nov 20;18(1):1140. doi: 10.1186/s12885-018-5052-8. PMID 30453906
- See also: Related Info — https://link-springer-com.udel.idm.oclc.org/article/10.1186/s12885-018-5052-8
- Available data/document: Study Protocol — https://link-springer-com.udel.idm.oclc.org/article/10.1186/s12885-018-5052-8